CLINICAL TRIAL: NCT01277315
Title: Open Safety and Tolerability Trial to Evaluate a Subcutaneous Injection Solution of 100 mg of Anakinra in Combination With Riluzol in Amyotrophic Lateral Sclerosis
Brief Title: Safety and Tolerability of Anakinra in Combination With Riluzol in Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Max Planck Institute for Infection Biology (Other)
Responsible Party: Principal Investigator, Thomas Meyer, MD, Prof. Dr. Thomas Meyer, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANA-ALS01
Record Dates: First submitted 2011-01-13; First posted 2011-01-14 (Estimated); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: ALS; Anakinra; Kineret; Progressive Muscular Atrophy; PMA; Safety Trial; Tolerability Trial
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Muscular Atrophy, Spinal | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Anakinra — Open Safety and Tolerability study to evaluate a subcutaneous application 100 mg of Anakinra in combination with Riluzol in Amyotrophic Lateral Sclerosis.

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) is an adult neurodegenerative disease that is caused by a selective degeneration of the motor nerve cells in the cortex and myelon. As a result of motor neurodegeneration, a progredient paralysis of the extremities and of the speaking, swallowing, and breathing musculature develops. ALS leads to death by respiratory insufficiency in a mean course of 3-5 years. So far, Riluzole is the only approved neuroprotective medication which effects a slight lifespan prolongation of 1.5 - 2.5 months. Riluzole inhibits the presynaptic glutamate release and lowers the level of glutamate liberated by activated microglia.

The researchers propose an investigational therapy of ALS with subcutaneous administration of 100 mg of Anakinra. The neuronal inflammation is a crucial pathogenetic factor of the motor neuron degeneration. Inflammatory processes are detectable in sporadic ALS, in the autosomal-dominant form of ALS and in transgenic mouse model. The rationale of this clinical trial is based on the anti-inflammatory effect of Anakinra. One of the key mediators of inflammatory response is Interleukin-1. Anakinra is a recombinant produced Interleukin-1 receptor antagonist. This gives Anakinra anti-inflammatory attributes that presumably reduce motor neuron degeneration and disease progression.

DETAILED DESCRIPTION:
Open Safety and Tolerability study to evaluate a subcutaneous application 100 mg of Anakinra in combination with Riluzol in Amyotrophic Lateral Sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 80 years of age
* Clinical diagnosis of amyotrophic lateral sclerosis with predominant affection of the lower motor neuron or the clinical ALS variant of progressive muscular atrophy (PMA)
* Clinical signs of lower motor neuron degeneration in at least one anatomic region beyond the brain stem
* Sporadic and familial ALS
* Onset of paresis six months to four years before study inclusion
* Treatment with riluzol 100mg/d at least 1 month before study inclusion

Exclusion Criteria:

* Diagnosis of amyotrophic lateral sclerosis with predominant affection or the upper motor neuron without clinical signs of a concurrent affection of the lower motor neuron in at least one anatomic region beyond the brain stem (spastic ALS) - Diagnosis of primary lateral sclerosis (PLS)
* Patients with known intolerance to anakinra, riluzol or one of the additives
* Clinically severe hypoventilation syndrome with vital capacity < 50%
* Pregnancy or breastfeeding
* Continuous non-invasive ventilation with ventilator-free time < 2 hours - Tracheotomy and mechanical ventilation
* Laboratory parameters outside the normal range that correspond to a clinically severe cardiovascular, pulmological, hematological, hepatological, metabolic or renal disease
* Malignancies
* Severe renal insufficiency (creatinine clearance < 30 ml/min)
* History of recurrent infections or a disease that may predispose to infections
* Severe neutropenia (absolute neutrophil count < 1.5 x 109/l)
* Monoclonal gammopathy of unknown significance
* Infections including infections with HIV and hepatitis B and C
* Dementia and unable to give informed consent
* History of epilepsy and epileptic seizures
* Contraindication to E coli-derived proteins, anakinra or any components of the product
* Concurrent therapy of anakinra and etanercept or other TNF blocking agents

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Number and Severity of adverse events (AE) | 1 month
Number and Severity of serious adverse events (SAE) | 1 month
Number and Severity of adverse drug reactions (ARD) | 1 month
Number and Severity of unexpected adverse drug reactions (UADR) | 1 month
Number and Severity of serious adverse drug reactions (SADR) | 1 month
Number and Severity of suspected unexpected serious adverse reaction (SUSAR) | 1 month
Pathological laboratory parameters | 1 month

SECONDARY OUTCOMES:
Long Term Tolerability and Safety of Anakinra in ALS Patients | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Meyer, MD, Principal Investigator — Charité University Hospital, Berlin, Germany
Locations (1):
- Charité University Hospital, Berlin, Germany

REFERENCES:
- [Derived] Maier A, Deigendesch N, Muller K, Weishaupt JH, Krannich A, Rohle R, Meissner F, Molawi K, Munch C, Holm T, Meyer R, Meyer T, Zychlinsky A. Interleukin-1 Antagonist Anakinra in Amyotrophic Lateral Sclerosis--A Pilot Study. PLoS One. 2015 Oct 7;10(10):e0139684. doi: 10.1371/journal.pone.0139684. eCollection 2015. PMID 26444282